CLINICAL TRIAL: NCT05758649
Title: Cardiovascular and Psychological Consequences of COVID-19
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: CE 2450
Record Dates: First submitted 2023-03-03; First posted 2023-03-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Post-COVID Conditions
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will assess cardiac and psychological profile at 2-3 months after recovery from COVID-19 infection.

DETAILED DESCRIPTION:
A significant proportion of patients hospitalized for COVID-19 showed laboratory signs of myocardial damage, detected by elevated troponin levels, and these were associated with more severe clinical course and higher mortality. Moreover, it is unknown how the health emergency and the associated conditions may have influenced and still influence the psychological experience of the affected people.

Thus, in order to promote continuity of care, post-COVID-19 disease clinics have therefore been activated dedicated to a specific follow-up program for monitoring long-term alterations and for the early identification of patients requiring rehabilitation.

The program includes a first follow-up visit (2-3 months after recovery) including cardiac (2D-echocardiography, six-minute walking test, autonomic function evaluation) and psychological (Patient Health Questionnaire-9 (PHQ-9) Generalized Anxiety Disorder-7 (GAD) National Stressful Events Survey PTSD Short Scale (NSESSS)) evaluation.

A second follow-up visit will be performed at 12 months in the form of structured interview,

ELIGIBILITY:
Inclusion Criteria:

* Recent discharge (≤ 3 months) from a COVID+ ward for SARS-CoV-2 disease

Exclusion Criteria:

* Serious clinical conditions (severe chronic inflammatory diseases, neoplasms, neurological pathologies).
* Non-Italian education, illiteracy, or return to illiteracy.
* Severe visual-perceptual deficits.
* Low motivation/interest or refusal to undergo the assessment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will refer to the disease clinics 2-3 months after discharge from the COVID-19 areas of ICS Maugeri.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
prevalence of patients with cardiovascular or psychological sequelae | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri, Pavia, Italy

REFERENCES:
- [Result] Vigore M, Steccanella A, Maffoni M, Torlaschi V, Gorini A, La Rovere MT, Maestri R, Bussotti M, Masnaghetti S, Fanfulla F, Pierobon A. Patients' Clinical and Psychological Status in Different COVID-19 Waves in Italy: A Quanti-Qualitative Study. Healthcare (Basel). 2023 Sep 6;11(18):2477. doi: 10.3390/healthcare11182477. PMID 37761674